CLINICAL TRIAL: NCT05315362
Title: Establishing Immunogenicity and Safety of Needle-free Intradermal Delivery by Solid Micro Needle Skin Patch of mRNA SARS-CoV-2 Vaccine as a Revaccination Strategy in Healthy Volunteers
Brief Title: Establishing Immunogenicity and Safety of Needle-free Intradermal Delivery of mRNA COVID-19 Vaccine
Acronym: MILESTONE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, aheroukens, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL80101.058.22
Record Dates: First submitted 2022-04-06; First posted 2022-04-07 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Vaccination; Infection; COVID-19
MeSH Terms: conditions — Infections; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: open-label, randomised-controlled, proof-of-concept vaccine study
Masking Description: only laboratory personnel is masked. Because of the different administration routes it is not possible to mask the participants or investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group - intradermal vaccination with patch (Experimental): Participants will receive 20 µg of mRNA-1273 vaccine through the intradermal route using a solid micro needle delivery system
  Interventions: Device: solid microneedle skin patch; Biological: mRNA-1273
- Control group - intramuscular vaccination with standard needle (Active Comparator): Participants will receive 20 µg of mRNA-1273 vaccine through the intramuscular route
  Interventions: Biological: mRNA-1273; Device: standard needle

INTERVENTIONS:
Device: solid microneedle skin patch — intradermal vaccination with a skin patch
  Arms: Intervention group - intradermal vaccination with patch
Biological: mRNA-1273 — administration of mRNA-1273 vaccine
Device: standard needle — intramuscular vaccination with a standard needle
  Arms: Control group - intramuscular vaccination with standard needle

SUMMARY:
COVID-19 vaccines are limited in supply, especially in low- and middle-income countries, leading to substantial morbidity and mortality. Despite the COVID-19 Vaccines Global Access (COVAX) Facility initiated by the WHO to provide vaccine access for low-income countries, probably 80% of the vaccine needs of participating countries will not be met soon.

In addition, there is an increasing demand for revaccination of the population globally, because of waning immunity which will further limit vaccine supplies. Exploring dose-sparing techniques, could therefore provide the solution to immunise more people with the same vaccine stockpile.

The intramuscular injection (IM) is the standard inoculation route of vaccines. However, the skin (dermis) is much richer in antigen presenting dendritic cells than muscle. As a consequence, a fractional vaccine dose introduced directly into the dermis (intradermal administration, ID) might be as effective as the intramuscular administration of the full standard dose to achieve a protective immune response. This principle has recently been demonstrated for the ID dermal delivery of one-fifth fractional dose mRNA-1273 (Spikevax, Moderna) vaccine.

However, needle-based immunisation has several limitations. Fear of needles makes immunisation a stressful event. In addition, needle stick injuries, as well as unsafe injection practices carry serious health risks. Therefore, the development of needle-free delivery has been identified as an important goal in global health care. The WHO reported that microneedle vaccine delivery is top priority and requires additional research to explore the benefits in more detail. A big advantage of intradermal delivery via a solid needle patch is not only the absence of needles and pain since no nerves are at the proximity where the needles are presented, but also the local delivery close to immune cells as with the above mentioned intradermal injection enables a much lower dose as compared to IM dosing. And since with the patch a larger skin surface is involved as compared to intradermal injection, even lower doses are possibly still immunogenic.

In this study, we will investigate the immunogenicity and safety in healthy volunteers of the needle-free intradermal delivery of a single fractional dose of 20µg mRNA-1273 LNP vaccine (Spikevax, Moderna) more than 3 months after primary vaccination with Comirnaty (Pfizer) vaccine and/or after having contracted COVID-19.

DETAILED DESCRIPTION:
Objectives Primary objective

* to describe immunogenicity and safety in healthy volunteers of the needle-free intradermal delivery of a single fractional dose of 20µg mRNA-1273 LNP vaccine (Spikevax, Moderna) more than 3 months after primary vaccination with Comirnaty (Pfizer) vaccine and/or after have contracted COVID-19.

Secondary objectives

* to describe the kinetics of the SARS-CoV-2 anti-Spike1 (S1) and Region Binding Domain (RBD) IgG binding antibodies elicited by needle-free intradermal or intramuscular delivery of mRNA-1273 vaccine in healthy volunteers after a single fractional dose of 20µg mRNA-1273 LNP vaccine
* to describe the kinetics of the SARS-CoV-2 neutralising antibodies elicited by needle-free intradermal or intramuscular delivery of mRNA-1273 vaccine in healthy volunteers after a single fractional dose of 20µg mRNA-1273 LNP vaccine

Exploratory objectives:

* to describe the kinetics of memory B-cell and plasma cell responses elicited by needle-free intradermal or intramuscular delivery of mRNA-1273 vaccine of a single fractional dose of 20µg mRNA-1273 LNP vaccine (Spikevax, Moderna)
* to describe the interferon-gamma release in whole blood in response to SARS-CoV 2 peptides after needle-free intradermal or intramuscular delivery of mRNA-1273 vaccine of a single fractional doses of 20µg mRNA-1273 LNP vaccine (Spikevax, Moderna)

Study design:

This is a Phase 2a, open-label, randomised-controlled, proof-of-concept vaccine study

Study population:

Healthy volunteers aged 18 - 40 years who have been vaccinated with Comirnaty (Pfizer) vaccine at least 3 months before

Intervention group:

Participants will receive 20 µg of mRNA-1273 vaccine through the needle-free intradermal route using a micro-needle delivery system.

Control group:

Participants will receive 20 µg of mRNA-1273 vaccine through the intramuscular route

Main study parameters/endpoints:

* Solicited local reactions and systemic events self-reported by diary on a daily basis over a 2-week period, telephone interview on D4, as well as by on site visits on D15 and D29
* Adverse events (AEs) until two weeks after administration
* Serious AEs (SAEs) until six months after administration
* Seroconversion for anti-spike IgG antibodies (D29)
* Geometric mean concentrations (GMC) for anti-spike IgG antibodies (D1, D29)

ELIGIBILITY:
Inclusion Criteria:

* Previously vaccinated with Comirnaty (Pfizer) and/or previously contracted COVID-19 at least 3 months before inclusion
* Healthy participants who are determined by medical history and clinical judgment of the investigator to be eligible for inclusion in the study. Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalisation for worsening disease during the 6 weeks before enrolment, can be included.
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Participants are willing to postpone their regular COVID-19 revaccination upon invitation by the municipal health center or general practitioner until four weeks after receiving the intervention (after the last sampling of D29).
* Capable of giving personal signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behaviour or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention(s).
* Receipt of medications intended to prevent COVID-19.
* Previous microbiological diagnosis of COVID-19.
* Previous COVID-19 vaccination other than Comirnaty (Pfizer)
* Individuals at high risk for severe COVID-19 (e.g. BMI > 40, diabetes, heart- end/or lung disease), who are planned to receive COVID vaccine within the next two months.
* Immunosuppressed individuals with known or suspected immunodeficiency, as determined by history.
* Individuals with an active autoimmune disease requiring therapeutic intervention.
* Receipt of systemic or topical corticosteroids.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Planned pregnancy within four weeks after injection.
* Positive serological test for SARS-CoV-2 anti-N IgM and/or IgG antibodies at screening visit.
* SARS-CoV-2 PCR-positive mid-turbinate/throat swab at the screening before receipt of the vaccine dose.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Receipt of any other non-study vaccine within 28 days, before receipt of the study dose.
* Anticipated receipt of any other non-study vaccine within 28 days, after the study dose administration.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2-spike protein-specific binding IgG antibody levels | 3 months
  SARS-CoV-2-spike protein-specific binding IgG antibody levels
adverse events | 1 month
  local and systemic reactions after intradermal vaccination with a solid microneedle patch

SECONDARY OUTCOMES:
SARS CoV 2 neutralizing antibody levels | 3 months
  SARS CoV 2 neutralizing antibody levels
Number of Spike-protein specific proliferating B-cells, plasma cells and B-memory cells | 6 months
  Number of Spike-protein specific proliferating B-cells, plasma cells and B-memory cells
INF-gamma concentration and other cytokine responses after over-night incubation | 3 months
  INF-gamma concentration and other cytokine responses after over-night incubation

CONTACTS AND LOCATIONS:
Overall Officials: Anna H Roukens, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prins MLM, Prins C, de Vries JJC, Visser LG, Roukens AHE. Establishing immunogenicity and safety of needle-free intradermal delivery by nanoporous ceramic skin patch of mRNA SARS-CoV-2 vaccine as a revaccination strategy in healthy volunteers. Virus Res. 2023 Sep;334:199175. doi: 10.1016/j.virusres.2023.199175. Epub 2023 Jul 21. PMID 37473964